CLINICAL TRIAL: NCT03091530
Title: Restoration of Glenohumeral Internal Rotation Deficit (GIRD) After Throwing: A Randomized Clinical Trail Comparing the Sleeper Stretch to the 90/90 Hip Lift With Balloon Blow Exercise
Brief Title: Glenohumeral Rotation After Throwing: RCT Comparing the Sleeper Stretch to the 90/90 Hip Lift With Balloon Blow Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00081964
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-01

CONDITIONS: Internal Rotation Contracture-shoulder
Keywords: Throwing; Sleeper Stretch; Balloon Blow; GIRD (Glenohumeral internal rotation deficit)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeper Stretch THEN Balloon Blow (Experimental): Sleeper Stretch CROSSOVER TO 90/90 Hip Lift with Balloon Blow Exercise
  Interventions: Other: Sleeper Stretch; Other: 90/90 Hip Lift with Balloon Blow Exercise
- Balloon Blow THEN Sleeper Stretch (Experimental): 90/90 Hip Lift with Balloon Blow Exercise CROSSOVER TO Sleeper Stretch
  Interventions: Other: Sleeper Stretch; Other: 90/90 Hip Lift with Balloon Blow Exercise

INTERVENTIONS:
Other: Sleeper Stretch — The sleeper stretch protocol will follow the process described by Wilk with the subject lying on his throwing shoulder side, with the lateral border of the scapula on the table, and the glenohumeral and elbow joints both at 90 degrees of flexion. Participants will be instructed to passively internally rotate the shoulder with gentle overpressure applied on the dorsum of the dominant arm wrist by the nondominant hand to the point of stretch on the posterior aspect of the shoulder. Stretches will be held for 20 seconds each and repeated 4 times for optimal sustained collagen elongation. This protocol will be performed on days 0-4 after the throwing session.
Other: 90/90 Hip Lift with Balloon Blow Exercise — The 90/90 Hip Lift with Balloon Blow Exercise (BBE) will follow the guidelines described by the Postural Restoration Institute. The subjects will lie supine with hips and knees flexed to 90 degrees, the right arm flexed to end range and resting on the floor. Using the left arm to hold the balloon, subjects will inhale fully and exhale into a balloon while holding a posterior pelvic tilt. The subjects inhale and then exhale into the balloon fully, then hold their breath for 5 seconds while putting their tongue on the roof of their mouth.

SUMMARY:
The primary purpose of this study is to determine if the loss of internal rotation following a throwing session is best restored through soft tissue stretching with the sleeper stretch or with scapular repositioning with the 90/90 hip lift with balloon blow exercise. This study will progress the body of research related to internal rotation deficits with regards to baseball throwers. The research will be relevant to clinicians who treat patients with baseball players with internal rotation loss.

High school baseball players will be the targeted subjects for this study. They will perform two exercises (one per week) designed to increase shoulder internal rotation over the course of three weeks with one week of rest between intervention weeks. The primary outcome will be shoulder internal rotation range of motion improvements over the course of one week's time. There are no known adverse risks to either intervention.

DETAILED DESCRIPTION:
Purpose of the Study: The primary purpose of this study is to determine if the loss of internal rotation following a throwing session is best restored through soft tissue stretching with the sleeper stretch or with scapular repositioning with the 90/90 hip lift with balloon blow exercise. This study will progress the body of research related to internal rotation deficits with regards to baseball throwers. The research will be relevant to clinicians who treat patients with baseball players with internal rotation loss.

Specific Aim: To determine if the glenohumeral internal rotation deficit (GIRD) is more effectively restored following a throwing session by performing the sleeper stretch (SS) or the 90/90 hip lift with balloon blow exercise (BBE).

Hypothesis: BBE will improve GIRD more effectively and quickly than the SS.

This is a prospective randomized trial comparing the efficacy of two exercises designed to improve shoulder internal rotation. Subjects meeting study criteria will be randomly allocated to each group as shown in the following CONSORT allocation diagram. Randomization will be performed via random number generator.

Each subject will participate in two week-long interventions with at least one week separating the two intervention weeks. During the week of intervention, the subject will have his baseline IR measured. He will then be instructed in how to perform a single exercise designed to improve internal rotation range of motion. Approximately half of the subjects will perform the Sleeper Stretch the first week, then the Balloon Blow Exercise the second week. The remaining group of subjects will perform the Balloon Blow Exercise during the first week, then the Sleeper Stretch the second week. Both exercises will be instructed by a physical therapist who commonly prescribes the exercises in the clinical setting. A written handout detailing the exercise instructions, frequency, and duration of the stretch will be provided for the subjects' reference (submitted with IRB application). The subject will perform this exercise throughout the week as directed by study personnel. Baseline measures of glenohumeral internal rotation (IR) with the shoulder positioned at 90 degrees of abduction in the scapular plane will be obtained using a goniometer, as described by Manske. These measurements will be repeated after the initiation of the intervention exercise at the following intervals: 2 hours, 1 day, 2 days, 3 days and 4 days. All measures of IR will be taken 3 times and the average of the three measures used in data analysis. The investigator performing the measures will be blinded to participant group assignment. When the subject completes both intervention weeks, he will be asked if he had a personal preference for either exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Active participation in competitive high school baseball at the time of study participation.
2. Ability to read, write, and speak the English language.

Exclusion Criteria:

1. Prior surgery to the dominant (throwing) shoulder
2. Any current upper extremity injury or limitation that restricts full participation in sport
3. Latex allergy secondary to use of latex material of the balloon
4. Any known inability to be physically present for daily testing during the weeks of the study

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-04-14 (Actual)

PRIMARY OUTCOMES:
Change In Shoulder Internal Rotation Range of Motion | baseline, 2 hours, 1 day, 2 days, 3 days, 4 days
  Goniometric measurement of passive shoulder internal rotation

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No